CLINICAL TRIAL: NCT02787525
Title: Comparison of Clinical Outcomes After Left Atrial Appendage Closure or Oral Anticoagulation in Patients With Atrial Fibrillation: A Retrospective Propensity Matched Study
Brief Title: Comparison of Outcomes After Left Atrial Appendage Closure or Oral Anticoagulation in Patients With Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-00630
Record Dates: First submitted 2016-05-25; First posted 2016-06-01 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: patients on anticoagulation: Questionnaire to patients with non-valvular atrial fibrillation on OAC or NOAC
  Interventions: Other: Questionnaire
- B: patients treated by LAA-Closure: Questionnaire to patient with non-valvular atrial fibrillation who underwent LAAC between 2009 and 2014 at the University hospitals Bern or Zurich
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A clinical sweep follow up will be performed in all patients of both groups and results will be analyzed. It will be in form of a standardized questionnaire and if necessary telephone interviews asking about thrombo-embolic events, stroke, death, any bleeding but also on their current medication, comorbidities (i.e. arterial hypertension, diabetes mellitus, renal impairment and liver disease), any hospitalizations and their quality of life. For all events, the source documents will be gathered from general physicians, cardiologists, hospitals or registry offices.
  The questionnaire will be sent by mail to the patients. If information is missing or unclear, patients and if necessary their treating physician will be contacted by phone.

SUMMARY:
The aim of the study is to compare intermedium-term clinical outcomes, including thromboembolic events and bleeding complications between patients with non-valvular atrial fibrillation treated with either oral anticoagulation or who had undergone LAA-closure (left atrial closure).

A questionnaire is sent to the patients and if there is some information missing or unclear, the investigators will contact the patient or the treating physicians to get the missing/unclear information.

The study population consists of 500 patients with non-valvular atrial fibrillation (AF) who underwent LAAC between the years 2009 and 2014 in two centers (the Bern University hospital und Zurich University hospital) and a similar group of 500 patients with non-valvular AF treated with oral anticoagulation (OAC).

In order to compare the two groups and reducing the bias due to confounding variables, a propensity score matching will be performed.

Study hypothesis is that left atrial appendage closure is non-inferior in terms of efficacy and safety in comparison to lifelong oral anticoagulation in patients with non-valvular atrial fibrillation.

DETAILED DESCRIPTION:
Non-valvular atrial fibrillation is the most common arrhythmia with an estimated prevalence of 1-2% in the general population, increasing with age. Patients with AF are at increased risk of thromboembolism, in particular ischemic stroke.

LAAC seems at the actual knowledge to be a valid alternative to OAC. The objective of this study is to compare intermedium-term clinical outcomes, including thromboembolic events and bleeding complications between patients receiving Amplatzer devices vs. propensity score matched patients treated with OAC.

A questionnaire is sent to the patients asking about thrombo-embolic events, stroke, death, any bleeding but also on their current medication, comorbidities (i.e. arterial hypertension, diabetes mellitus, renal impairment and liver disease), any hospitalizations and their quality of life. If there is some information missing or unclear, the investigators will contact the patient or the treating physicians to get the missing information.

The study is an investigator-initiated, retrospective analysis of prospectively collected data. The study population consists of 500 patients with non-valvular AF who underwent LAAC between the years 2009 and 2014 in two centers (the Bern University hospital und Zurich University hospital) and a propensity score matched patients group of 500 patients with non-valvular AF treated with OAC.

Covariates for matching will be age, gender, renal function, coronary artery disease and its status of revascularization, left-ventricular function, HAS-BLED and CHA2DS2-VASc-Score.

Study hypothesis is that left atrial appendage closure is non-inferior in terms of efficacy and safety in comparison to lifelong oral anticoagulation in patients with non-valvular atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Written informed consent to participate in the study
* Paroxysmal, persistent, or permanent non-valvular atrial fibrillation.
* Group A ("OAC"): Having been hospitalized between 2009 and 2014 in the Bern university hospital and discharged with either OAC or NOAC.
* Group B (LAA-closure): Underwent LAAC between 2009 and 2014 at the University hospitals Bern or Zurich

Exclusion Criteria:

* No full data on matching criteria (which are described below under "study design")
* Only for group A: Not matched patients having been dropped out after the propensity score matching

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Group A ("OAC"): Patients having been hospitalized between 2009 and 2014 in the Bern university hospital and discharged with either OAC or NOAC.
  * Group B (LAA-closure): Patients who underwent LAAC between 2009 and 2014 at the University hospitals Bern or Zurich
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2016-07; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of intermedium-term clinical outcomes, including thromboembolic events and bleeding complications in patients receiving Amplatzer devices vs. propensity score matched patients treated with OAC. | Clinical sweep follow up, the mean follow-up will be approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Gloeckler, PD Dr. med, Principal Investigator — University hospital Berne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reddy VY, Sievert H, Halperin J, Doshi SK, Buchbinder M, Neuzil P, Huber K, Whisenant B, Kar S, Swarup V, Gordon N, Holmes D; PROTECT AF Steering Committee and Investigators. Percutaneous left atrial appendage closure vs warfarin for atrial fibrillation: a randomized clinical trial. JAMA. 2014 Nov 19;312(19):1988-98. doi: 10.1001/jama.2014.15192. PMID 25399274
- [Background] Reddy VY, Mobius-Winkler S, Miller MA, Neuzil P, Schuler G, Wiebe J, Sick P, Sievert H. Left atrial appendage closure with the Watchman device in patients with a contraindication for oral anticoagulation: the ASAP study (ASA Plavix Feasibility Study With Watchman Left Atrial Appendage Closure Technology). J Am Coll Cardiol. 2013 Jun 25;61(25):2551-6. doi: 10.1016/j.jacc.2013.03.035. Epub 2013 Apr 10. PMID 23583249
- [Background] Tzikas A, Shakir S, Gafoor S, Omran H, Berti S, Santoro G, Kefer J, Landmesser U, Nielsen-Kudsk JE, Cruz-Gonzalez I, Sievert H, Tichelbacker T, Kanagaratnam P, Nietlispach F, Aminian A, Kasch F, Freixa X, Danna P, Rezzaghi M, Vermeersch P, Stock F, Stolcova M, Costa M, Ibrahim R, Schillinger W, Meier B, Park JW. Left atrial appendage occlusion for stroke prevention in atrial fibrillation: multicentre experience with the AMPLATZER Cardiac Plug. EuroIntervention. 2016 Feb;11(10):1170-9. doi: 10.4244/EIJY15M01_06. PMID 25604089
- [Background] Nietlispach F, Gloekler S, Krause R, Shakir S, Schmid M, Khattab AA, Wenaweser P, Windecker S, Meier B. Amplatzer left atrial appendage occlusion: single center 10-year experience. Catheter Cardiovasc Interv. 2013 Aug 1;82(2):283-9. doi: 10.1002/ccd.24872. Epub 2013 Mar 22. PMID 23412815